CLINICAL TRIAL: NCT00767156
Title: Subjective and Instrumental Evaluation of the Effects of Treatments With Two Sea Buckthorn Oil Products on Cutaneous Aging
Brief Title: Effects of Oral and Topical Sea Buckthorn Oil Treatments on Skin Aging
Acronym: SBanti-aging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Skin and Product Evaluation, Italy (Other)
Collaborators: Aromtech Ltd. (Industry)
Responsible Party: Adriana Bonfigli, ISPE
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E11UE15UE25US14C
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-10

CONDITIONS: Skin Aging
Keywords: Sea buckthorn oil, Oral and topical treatment, Skin aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- SBA24 capsule plus Omega7 cream (Active Comparator): the subjects took SBA24 sea buckthorn oil capsule and apply Omega7 cream
  Interventions: Dietary Supplement: SBA24 Sea Buckthorn Oil Capsule
- SBA24 capsule plus base cream (Active Comparator): the subjects took SBA24 sea buckthorn oil capsule and apply a base cream
  Interventions: Dietary Supplement: SBA24 Sea Buckthorn Oil Capsule
- Omega7 Cream (Active Comparator): The subjects Omega 7 Sea Buckthorn Oil Cream, twice per day
  Interventions: Other: Omega7 Sea Buckthorn Oil Cream
- Base cream (Placebo Comparator): The subjects use base cream on the face, twice per day
  Interventions: Other: Base cream

INTERVENTIONS:
Other: Omega7 Sea Buckthorn Oil Cream — The subjects use Omega7 Sea Buckthorn Oil Cream on the face, twice per day
  Arms: Omega7 Cream
Other: Base cream — The subjects use the base cream on the face, twice per day
  Arms: Base cream
Dietary Supplement: SBA24 Sea Buckthorn Oil Capsule — The subjects take SBA24 sea Buckthorn Oil Capsules, 2 x 2 capsules (2.0 g oil) per day and use topically Omega7 Sea Buckthorn Oil Cream, twice per day.
  Other Names: Omega7/Membrasin Capsule, Omega7 Cream
  Arms: SBA24 capsule plus Omega7 cream
Dietary Supplement: SBA24 Sea Buckthorn Oil Capsule — Teh subjects took SBA24 Sea Buckthorn Oil Capsule, 2 x 2 capsules (2 g oil) per day and use topically the base cream, twice per day
  Other Names: Omega7/Membrasin/SBA24 Sea Buckthorn Oil Capsule
  Arms: SBA24 capsule plus base cream

SUMMARY:
The effect of oral supplementation of SBA24 sea buckthorn oil capsule and topical application of Omega7 sea buckthorn cream on skin ageing is studied in a single blind, parallel study.

DETAILED DESCRIPTION:
The study is carried out on two groups of female volunteers, 30 in each group, of age 30 to 60 years, in compliance with the principles established by the World Medical Association in the Declaration of Helsinki. In group I, the subjects took SBA24 sea buckthorn oil capsule (2 x 2 capsules per day) and apply two different creams on the face, one cream on each half of the face, twice per day. In group II, the subjects apply only the two creams, one cream on each half of the face, twice per day, for 8 weeks.

The assessment is performed on the skin surface of the periocular areas.

The efficacy of the active products is assessed on the skin face at the beginning, after 4 weeks and after 8 weeks of treatment using the following instrumental measurements:

* cutaneous elasticity (CUTOMETER SEM 575 Courage & Khazaka);
* cutaneous hydration level (CORNEOMETER CM 825 Combi 3 Courage & Khazaka);
* cutaneous roughness by cutaneous replicas and image analysis (Quantilines, Monaderm); Determination of benefit is based on instrumental measurements and subject self-assessment questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects 30 - 60 years old with Fitzpatrick skin type I-IV & in good general health, with facial skin manifestation related to photoaging (wrinkles, dyschromias, tissue looseness etc.)
* Subjects must have discontinued the use of topical retinoid products for 6 months prior to study entry and of systemic retinoids for 1 year prior to study entry.
* Subjects must have discontinued the use of topical alpha-hydroxy, &/or beta-hydroxy products for 45 days prior to study entry & all other topical facial medication to the skin immediately prior to study entry.
* Subjects must have discontinued the use of systemic antiaging or antioxidant products for at least 2 months prior to study entry.
* Subjects must be willing & able to follow all study directions & to commit to all follow-up visits for the duration of the study.
* Subjects must have completed the informed consent process.
* Subjects must be willing to avoid direct daily sun exposure on the face or the use of tanning beds.

Exclusion Criteria:

* Pregnant or nursing females.
* Subjects with a history of unusual skin reactions to skin care toiletry products, cosmetics, or sensitivity to any of the test article components.
* Previous facial treatments with any dermal fillers (i.e. collagen, hyaluronic acid etc)
* Concurrent therapy, systemic diseases, or skin disorders (such as eczema, psoriasis, severe acne etc.) which may interfere with the evaluation of the test articles or increase risk to the subject.
* Subjects currently involved in another clinical investigation or who have been involved within a period of 30 days prior to admission in this study.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-11 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Decrease of signs of skin aging | 8 weeks

SECONDARY OUTCOMES:
Subjects self-assessment of the efficacy of the treatment | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Bonfigli, PhD, Principal Investigator — Research Director
Locations (1):
- ISPE Srl, Milan, Italy